CLINICAL TRIAL: NCT00787072
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of AZD8075 in Healthy Male Volunteers
Brief Title: AZD8075 Single Ascending Dose Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After reports of turbidity in urine in 4 of 8 volunteers in the 4th cohort, the study was halted temporarily.
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist, Medical Science Director, AstraZeneca R&D Lund, Sweden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3801C00001
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8075
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8075 — Single dose, the starting dose will be 7 mg, oral suspension, with up to 8 dose escalations not exceeding AstraZeneca pre-defined upper exposure limits.
  Arms: 1
Drug: Placebo — Oral suspension
  Arms: 2

SUMMARY:
The aim of this study is to assess the safety, tolerability and pharmacokinetics of single ascending oral doses of AZD8075 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures.
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg.
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start.

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the result of the study, or the subject's ability to participate
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs (vital signs (ie, supine BP and pulse) or ECG at baseline, which, in the opinion of the investigator, may put the subject at risk.
* Participation in another investigational drug study within 3 months before Visit 2 or participation in a method development study (no drug) 1 month prior to Visit 2

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | Frequent sampling occasions during study days

SECONDARY OUTCOMES:
PK variables | Frequent sampling occasions during study days

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Wolfgang Kühn, Principal Investigator — Quintiles, Uppsala, Sweden
Locations (1):
- Research Site, Uppsala, Sweden